CLINICAL TRIAL: NCT04916470
Title: Effect of Semaglutide 2.4 mg Once-weekly on Function and Symptoms in Subjects With Obesity-related Heart Failure With Preserved Ejection Fraction, and Type 2 Diabetes
Brief Title: Research Study to Look at How Well Semaglutide Works in People Living With Heart Failure, Obesity and Type 2 Diabetes
Acronym: STEP HFpEF DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX9536-4773; U1111-1257-5069 (Other: World Health Organization (WHO)); 2020-004170-22 (EudraCT Number)
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF) and Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide 2.4 mg once weekly (OW) (Experimental): Participants will receive semaglutide injections for 52 weeks.
  Interventions: Drug: Semaglutide
- Semaglutide placebo OW (Placebo Comparator): Participants will receive semaglutide placebo injections for 52 weeks.
  Interventions: Drug: Placebo (Semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Participants will receive semaglutide subcutaneous (s.c.; under the skin) injection(s) once-weekly for 52 weeks. Dose will be gradually increased to 2.4 mg: 0.25 mg from week 1 to 4, 0.5 mg from week 5 to 8, 1.0 mg from week 9 to 12, 1.7 mg from week 13 to 16 and 2.4 mg from week 17 to week 52.
  Arms: Semaglutide 2.4 mg once weekly (OW)
Drug: Placebo (Semaglutide) — Participants will receive semaglutide matching placebo s.c. injection(s) once-weekly for 52 weeks.
  Arms: Semaglutide placebo OW

SUMMARY:
This study will look at how participants' daily life is affected by their heart failure. The study will also look at the change in participants' body weight.

This study will compare the effect of semaglutide (a new medicine) compared to "dummy" medicine on body weight and heart failure symptoms.

Participants will either get semaglutide or "dummy" medicine, which treatment participants get is decided by chance.

Participants will need to take 1 injection once a week. The study medicine is injected with a thin needle in a skin fold in the stomach area, thigh or upper arm.

During the study participants will have talks with the study staff about healthy lifestyle and physical activity.

The study will last for about 59 weeks, that is a little more than 1 year. Participants will have 12 clinic visits with the study doctor.

* At 6 of the visits participants will have blood samples taken.
* At 5 of the visits participants will be asked to fill in a questionnaire
* At 4 of the visits participants will have to do a 6-minute walking test
* At 3 of the visits participants will have a test to check the heart.
* participants will have their eyes checked before or at the start of the study and at the end of the study

Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Body mass index (BMI) greater than or equal to 30.0 kg/m^2
* New York Heart Association (NYHA) Class II-IV
* Left ventricular ejection fraction (LVEF) greater than or equal to 45% at screening
* Diagnosed with T2D greater than or equal to 90 days prior to the day of screening
* HbA1c of below or equal to 10.0% as measured at the screening visit

Exclusion Criteria:

* A self-reported change in body weight greater than 5 kg (11 lbs) within 90 days before screening irrespective of medical records
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Change in KCCQ (Kansas City Cardiomyopathy Questionnaire) clinical summary score | From baseline (week 0) to end of treatment (week 52)
  Score on a scale of 0 to 100 where the score 100 means the least burden for the participant.
Change in body weight | From baseline (week 0) to end of treatment (week 52)
  Percentage (%)

SECONDARY OUTCOMES:
Change in 6-minute walking distance | From baseline (week 0) to end of treatment (week 52)
  Measured in metres
Hierarchical composite of time to all-cause death | From baseline (week 0) to end of study (week 57)
  Measured as total wins for each treatment group.
Hierarchical composite of number of heart failure events requiring hospitalisation or urgent heart failure visit | From baseline (week 0) to end of study (week 57)
  Measured as total wins for each treatment group
Hierarchical composite of time to first heart failure event requiring hospitalisation or urgent heart failure visit | From baseline (week 0) to end of study (week 57)
  Measured as total wins for each treatment group.
Hierarchical composite of difference at least 15 inKansas City Cardiomyopathy Questionnaire (KCCQ) clinical summary score change from baseline to 52 weeks | From baseline (week 0) to end of study (week 57)
  Measured as total wins for each treatment group.
Hierarchical composite of difference at least 10 in KCCQ clinical summary score change from baseline to 52 weeks | From baseline (week 0) to end of study (week 57)
  Measured as total wins for each treatment group.
Hierarchical composite of difference at least 5 in KCCQ clinical summary score change from baseline to 52 weeks | From baseline (week 0) to end of study (week 57)
  Measured as total wins for each treatment group.
Hierarchical composite of difference at least 30 metres in six-minute walking distance change from baseline to 52 weeks (assessed by the win ratio) | From baseline (week 0) to end of study (week 57)
  Measured as total wins for each treatment group.
Change in C-Reactive Protein | From baseline (week -2) to end of treatment (week 52)
  Presented as ratio to baseline
Participant achieving 10% weight loss or more (Yes/No) | From baseline (week 0) to end of treatment (week 52)
  Count of participants
Participant achieving 15% weight loss or more (Yes/No) | From baseline (week 0) to end of treatment (week 52)
  Count of participants
Participant achieving 20% weight loss or more (Yes/No) | From baseline (week 0) to end of treatment (week 52)
  Count of participants
Participant improving 5 points or more in KCCQ clinical summary score | From baseline (week 0) to end of treatment (week 52)
  Count of participants
Participant improving 10 points or more in KCCQ clinical summary score (Yes/No) | From baseline (week 0) to end of treatment (week 52)
  Count of participants
Change in KCCQ overall summary score | From baseline (week 0) to end of treatment (week 52)
  Score on a scale of 0 to 100 where the score 100 means the least burden for the participant.
Participant achieving threshold for clinically meaningful within-subject change in KCCQ-CSS | From baseline (week 0) to end of treatment (week 52)
  Count of participants
Participant achieving threshold for clinically meaningful within-subject change in 6MWD | From baseline (week 0) to end of treatment (week 52)
  Count of participants
Change in waist circumference | From baseline (week 0) to end of treatment (visit 52)
  Measured in centimetre (cm)
Change in systolic blood pressure | From baseline (week -2) to end of treatment (week 52)
  Measured in millimetre of mercury (mmHg)
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 52)
  Measured in percentage (%)-point
Number of treatment emergent severe or clinically significant hypoglycaemia episodes | From baseline (week 0) to end of trial (week 57)
  Count of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (Dept.1452), Study Director — Novo Nordisk A/S
Locations (176):
- United States (53):
  - Eastern Shore Rsrch Inst, LLC, Fairhope, Alabama
  - Mobile Heart Specialists, Mobile, Alabama
  - National Heart Institute Cal, Beverly Hills, California
  - John Muir Physicians Network, Concord, California
  - Valley Clinical Trials, Covina, California
  - Keck Medical Center of USC - Outpatient Clinic, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Lundquist Inst-Biomed Innovtn, Torrance, California
  - New West Physicians,Inc., Golden, Colorado
  - Excel Med Ctr Clinical Trials, Boca Raton, Florida
  - Bay Area Cardiology Associates, P.A., Brandon, Florida
  - Baptist Heart Specialists_Jacksonville, Jacksonville, Florida
  - CV Res Ctr of S Florida, Miami, Florida
  - Endeavor Health Clinical Operations-NCH, Arlington Heights, Illinois
  - Endeavor Health Glenbook Hosp, Evanston, Illinois
  - Northwestern University_Chicago_0, Evanston, Illinois
  - Chicago Medical Research LLC, Hazel Crest, Illinois
  - Deaconess Specialty Physicians, Evansville, Indiana
  - Ascension St. Vincent Medical Group, Indianapolis, Indiana
  - Cardiovascular Rsrch of NW_IN, Munster, Indiana
  - Cotton-O'Neil Heart Center, Topeka, Kansas
  - Baptist Health Woodland, Elizabethtown, Kentucky
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Grace Research, LLC, Bossier City, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Clinical Trials of Ame, LLC, Monroe, Louisiana
  - Grace Research, LLC_Shreveport, Shreveport, Louisiana
  - Louisiana Heart Center_Slidell, Slidell, Louisiana
  - Ascension Saint Agnes Heart Ca, Baltimore, Maryland
  - MedStar Good Samaritan Hosp, Baltimore, Maryland
  - John Hopkins Hospital, Baltimore, Maryland
  - Elite Research Center, Flint, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - St Louis Heart & Vascular, P.C., St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - CHI Health Clinic Cardiology (CUMC - Bergan Mercy), Omaha, Nebraska
  - St Francis Hospital Lindner Research Center, Greenvale, New York
  - NY Presbyt Hosp-W Cornell Med, New York, New York
  - Carteret Medical Group, Morehead City, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Lindner Center,Christ Hospital, Cincinnati, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Sanford Health_Sioux Falls, Sioux Falls, South Dakota
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Angio Cardiac Care of Texas, Houston, Texas
  - Cardiology Consultants of Danville Inc., Danville, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Argentina (8):
  - CEMEDIC, CABA, Buenos Aires
  - Centro de Investigación y Prevención Cardiovascular, CABA
  - CEMEDIC, CABA
  - Cardiología Palermo Duplicate, Ciudad Autónoma de Buenos Aire
  - Cardiología Palermo, Ciudad Autónoma de Buenos Aire
  - Instituto de Cardiología de Corrientes, Corrientes
  - Consultorio Integral de Atención al Diabético, Morón
  - Sanatorio Britanico S.A., Rosario, Santa Fe
- Austria (8):
  - Krankenhaus St. Josef Braunau, Braunau am Inn
  - Medizinische Universität Graz, Graz
  - Fließer-Görzer [Ordination], Saint Stefan
  - Medizinische Universität Wien, Vienna
  - Klinik Favoriten, Vienna
  - Imed 19- privat, Vienna
  - AKH Universitätsklinik für Innere Medizin II, Vienna
  - Universitätsklinik für Innere Medizin II, Vienna
- Canada (14):
  - University of Calgary_Calgary, Calgary, Alberta
  - Univ of Alberta Hosp Edmonton, Edmonton, Alberta
  - North Shore Heart Centre, North Vancouver, British Columbia
  - SMH Cardiology Clinical Trials Inc., Surrey, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Partnrs Adv Cardio Eval (PACE), Newmarket, Ontario
  - Oakville Cardiovascular Research LP, Oakville, Ontario
  - Heart Health Institute Research, Inc., Scarborough Village, Ontario
  - Dr. Louis Yao, Weston, Ontario
  - ViaCar Recherche Clinique Inc, Brossard, Quebec
  - Applied Med Inf Res, Montreal, Quebec
  - Ctr de Med Metab de Lanaudiere, Terrebonne, Quebec
  - Institut universitaire de cardiologie, Québec
- Czechia (5):
  - Edumed Broumov, Broumov
  - Fakultní poliklinika VFN ambulance Srdecniho selhani, Prague
  - IKEM, Prague
  - MEDICON a.s., Prague
  - Poliklinika Holešovice VISIONARY - Medicon Pharm s.r.o., Prague
- Germany (10):
  - Charité - Campus Virchow-Klinikum - Kardiologie, Angiologie und Intensivmedizin (CRU), Berlin
  - Cardiologicum Dresden und Pirna - MVZ "Am Felsenkeller" (Dresden), Dresden
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt
  - Medical Center - University Of Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Freiburg - Medical Center, Freiburg im Breisgau
  - B. Braun Ambulantes Herzzentrum Kassel MVZ GmbH, Kassel
  - Universitätsklinikum Leipzig - Klinik und Poliklinik für Kardiologie, Leipzig
  - Universitätsmedizin Mainz, Kardiologie I, Studienzentrum, Mainz
  - Universitatsklinikum Würzburg - Zentrum für Herzinsuffizienz, Würzburg
- Hungary (10):
  - Lausmed Kft., Baja, Bács-Kiskun county
  - Selye János Kórház, Komárom, Komárom-Esztergom
  - Szent Margit Rendelőintézet Nonprofit Kft., Budapest
  - Semmelweis Egyetem Szent Rókus Klinikai Tömb, Budapest
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Semmelweis Egyetem Városmajori Szív- és Érgyógyászat, Budapest
  - Jahn Ferenc Dél-pesti Kórház és Rendelőintézet, Budapest
  - DE KK Kardiológiai és Szívsebészeti klinika, Debrecen
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház, Miskolc
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg
- India (19):
  - Krishna Institute of medical sciences Ltd, Secunderabad, A.P.
  - CIMS- Care Institute of Medical Sciences, Ahmedabad, Gujarat
  - Rhythm Heart Institute, Vadodara, Gujarat
  - K R Hospital, Mysore, Karnataka
  - Lisie Hospital, Kochi, Kerala
  - Vijan Cardiac & Critical Care, Nashik, Maharashtra
  - Vijan Hospital & Research Centre, Nashik, Maharashtra
  - G B Pant Institute of Postgraduate Medical Education and Research, New Delhi, National Capital Territory of Delhi
  - Max Super Speciality Hospital, Saket, New Delhi, National Capital Territory of Delhi
  - Batra Hospital and Medical Research Center, New Delhi, National Capital Territory of Delhi
  - VMMC & Safdarjung Hospital, New Dehli, New Delhi
  - SP Medical College & A.G.Hospital Bikaner, Bikaner, Rajasthan
  - SP Medical College, Bikaner, Rajasthan
  - Apollo Hospitals Education & Research Foundation, Chennai, Tamil Nadu
  - Gandhi Memorial Hospital- King George's Medical University, Lucknow, Uttar Pradesh
  - G B Pant Institute of Postgraduate Medical Education and Res, New Delhi
  - Dr. BL Kapur Memorial Hospital, New Delhi
  - Max Super Speciality Hospital_New Delhi, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
- Israel (5):
  - Hadassah Ein Karam MC - Cardio Department, Jerusalem
  - Western Galilee MC - Cardiology Department, Nahariya
  - Rabin MC Beilinson - Heart Failure Unit, Petah Tikva
  - Sourasky MC - Cardio Vascular Research Center, Tel Aviv
  - Sheba MC - Cardiology Clinical Research Unit, Tel Litwinsky
- Italy (7):
  - Spedali Civili Brescia, Brescia, Bs
  - A.O.U. Ferrara, Sant'Anna, Cona (Ferrara), Fe
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo, Lombardy
  - Centro Cardiologico Monzino, Milan
  - Azienda Ospedaliera di Padova - MASTER, Padua
  - A.O.U. Policlinico Umberto I, Roma
  - Policlinico A. Gemelli IRCCS, Rome
- Japan (8):
  - Hyogo Prefectural HarimaHimeji General Medical Center_Cardiology, Himeji-shi, Hyogo
  - Kokura Memorial Hospital_Cardiology, Kitakyushu-shi,Fukuoka
  - Okayama University Hospital_Cardiovascular Medicine, Okayama-shi, Okayama
  - Omihachiman Community Medical Center_Omihachiman-shi, Siga, Omihachiman-shi, Siga
  - Osaka City General Hospital_Endocrinology and Diabetes Mellitus, Osaka
  - Medical Research Institute KITANO HOSPITAL_Cardiovascular Medicine, Osaka-shi, Osaka
  - Hanaoka Seishu Memorial Hosp._Cardiovascular Medicine, Sapporo-shi, Hokkaido
  - Tokyo Shinagawa Hospital_Cardiovascular Medicine, Tokyo
- Netherlands (7):
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Rode Kruis Ziekenhuis Beverwijk, Beverwijk
  - UMC Groningen, Groningen
  - Saxenburgh Medisch Centrum, Hardenberg
  - Frisius MC Leeuwarden, Leeuwarden
  - Bravis Ziekenhuis, Roosendaal
- Poland (6):
  - Malopolskie Centrum Sercowo-Naczyniowe, Chrzanów, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku K. Kardio, Bialystok, Podlaskie Voivodeship
  - Ind. Prak. Lek. w dziedz. Kardiologii lek. med. K. Cymerman, Gdynia, Pomeranian Voivodeship
  - Pro Familia Altera Sp. z o.o., Katowice, Silesian Voivodeship
  - I Katedra i Klinika Kardiologii WUM SPCSK, Warsaw
  - Uniwersytecki Szpital Kliniczny nr 2 Uniwersytetu Medycznego w Łodzi, Lodz, Łódź Voivodeship
- Spain (3):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Clínica Nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (3):
  - Dept of Med Sahlgrenska/Östra, Gothenburg
  - Medicinkliniken Ryhov, Jönköping
  - Hjärtmottagningen, Uppsala
- United Kingdom (10):
  - Ninewells Hospital, Dundee
  - Glasgow Clinical Research Facility, Glasgow
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Wycombe General Hospital, High Wycombe
  - Aintree University Hospital, Liverpool
  - University Hospital Aintree, Liverpool
  - Manchester Royal Infirmary_Manchester_0, Manchester
  - Manchester Royal Infirmary, Manchester
  - Great Western Hospital, Swindon

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Kosiborod MN, Abildstrom SZ, Borlaug BA, Butler J, Christensen L, Davies M, Hovingh KG, Kitzman DW, Lindegaard ML, Moller DV, Shah SJ, Treppendahl MB, Verma S, Petrie MC. Design and Baseline Characteristics of STEP-HFpEF Program Evaluating Semaglutide in Patients With Obesity HFpEF Phenotype. JACC Heart Fail. 2023 Aug;11(8 Pt 1):1000-1010. doi: 10.1016/j.jchf.2023.05.010. Epub 2023 May 21. PMID 37294245
- [Derived] Borlaug BA, Kitzman DW, Patel S, Chinnakondepalli KM, Butler J, Davies MJ, Petrie MC, Shah SJ, Verma S, Nunez J, Einfeldt MN, Liisberg K, Salsali A, Kosiborod MN; STEP-HFpEF Trial Committees and Investigators. Semaglutide and Exercise Function in Obesity-Related HFpEF: Insights From the STEP-HFpEF Program. JACC Heart Fail. 2025 Nov;13(11):102660. doi: 10.1016/j.jchf.2025.102660. Epub 2025 Oct 3. PMID 41045908
- [Derived] Pandey A, Kitzman DW, Chinnakondepalli KM, Patel S, Borlaug BA, Butler J, Davies MJ, Shah SJ, Verma S, Ronnback C, Domdey A, Liisberg K, Schou M, Perna E, Ahmed FZ, Fu M, Petrie MC, Kosiborod MN. Frailty and Effects of Semaglutide in Obesity-Related HFpEF: Findings From the STEP-HFpEF Program. JACC Heart Fail. 2025 Oct;13(10):102610. doi: 10.1016/j.jchf.2025.102610. Epub 2025 Sep 15. PMID 40956259
- [Derived] Davies MJ, van der Meer P, Verma S, Patel S, Chinnakondepalli KM, Borlaug BA, Butler J, Kitzman DW, Shah SJ, Harring S, Salsali A, Rasmussen S, von Lewinski D, Abhayaratna W, Petrie MC, Kosiborod MN; STEP-HFpEF Trials Committees and Investigators. Semaglutide in obesity-related heart failure with preserved ejection fraction and type 2 diabetes across baseline HbA1c levels (STEP-HFpEF DM): a prespecified analysis of heart failure and metabolic outcomes from a randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2025 Mar;13(3):196-209. doi: 10.1016/S2213-8587(24)00304-8. Epub 2025 Jan 20. PMID 39848268
- [Derived] Kosiborod MN, Deanfield J, Pratley R, Borlaug BA, Butler J, Davies MJ, Emerson SS, Kahn SE, Kitzman DW, Lingvay I, Mahaffey KW, Petrie MC, Plutzky J, Rasmussen S, Ronnback C, Shah SJ, Verma S, Weeke PE, Lincoff AM; SELECT, FLOW, STEP-HFpEF, and STEP-HFpEF DM Trial Committees and Investigators. Semaglutide versus placebo in patients with heart failure and mildly reduced or preserved ejection fraction: a pooled analysis of the SELECT, FLOW, STEP-HFpEF, and STEP-HFpEF DM randomised trials. Lancet. 2024 Sep 7;404(10456):949-961. doi: 10.1016/S0140-6736(24)01643-X. Epub 2024 Aug 30. PMID 39222642
- [Derived] Solomon SD, Ostrominski JW, Wang X, Shah SJ, Borlaug BA, Butler J, Davies MJ, Kitzman DW, Verma S, Abildstrom SZ, Nygaard Einfeldt M, Rasmussen S, Abhayaratna WP, Ahmed FZ, Ben-Gal T, Chopra V, Ito H, Merkely B, Nunez J, Senni M, van der Meer P, Wolf D, Petrie MC, Kosiborod MN; STEP-HFpEF Trial Committees and Investigators. Effect of Semaglutide on Cardiac Structure and Function in Patients With Obesity-Related Heart Failure. J Am Coll Cardiol. 2024 Oct 22;84(17):1587-1602. doi: 10.1016/j.jacc.2024.08.021. Epub 2024 Aug 30. PMID 39217567
- [Derived] Verma S, Butler J, Borlaug BA, Davies MJ, Kitzman DW, Petrie MC, Shah SJ, Jensen TJ, Rasmussen S, Ronnback C, Merkely B, O'Keefe E, Kosiborod MN; STEP-HFpEF and STEP-HFpEF DM Investigators. Atrial Fibrillation and Semaglutide Effects in Obesity-Related Heart Failure With Preserved Ejection Fraction: STEP-HFpEF Program. J Am Coll Cardiol. 2024 Oct 22;84(17):1603-1614. doi: 10.1016/j.jacc.2024.08.023. Epub 2024 Aug 30. PMID 39217565
- [Derived] Verma S, Petrie MC, Borlaug BA, Butler J, Davies MJ, Kitzman DW, Shah SJ, Ronnback C, Abildstrom SZ, Liisberg K, Wolf D, von Lewinski D, Lelonek M, Melenovsky V, Senni M, Kosiborod MN; STEP-HFpEF Trial Committees and Investigators. Inflammation in Obesity-Related HFpEF: The STEP-HFpEF Program. J Am Coll Cardiol. 2024 Oct 22;84(17):1646-1662. doi: 10.1016/j.jacc.2024.08.028. Epub 2024 Aug 30. PMID 39217564
- [Derived] Schou M, Petrie MC, Borlaug BA, Butler J, Davies MJ, Kitzman DW, Shah SJ, Verma S, Patel S, Chinnakondepalli KM, Harring S, Abildstrom SZ, Liisberg K, Kosiborod MN; STEP-HFpEF Trial Committees and Investigators. Semaglutide and NYHA Functional Class in Obesity-Related Heart Failure With Preserved Ejection Fraction: The STEP-HFpEF Program. J Am Coll Cardiol. 2024 Jul 16;84(3):247-257. doi: 10.1016/j.jacc.2024.04.038. Epub 2024 Jun 23. PMID 38913004
- [Derived] Verma S, Butler J, Borlaug BA, Davies M, Kitzman DW, Shah SJ, Petrie MC, Barros E, Ronnback C, Vestergaard LS, Schou M, Ezekowitz JA, Sharma K, Patel S, Chinnakondepalli KM, Kosiborod MN; STEP-HFpEF Trial Committees and Investigators. Efficacy of Semaglutide by Sex in Obesity-Related Heart Failure With Preserved Ejection Fraction: STEP-HFpEF Trials. J Am Coll Cardiol. 2024 Aug 27;84(9):773-785. doi: 10.1016/j.jacc.2024.06.001. Epub 2024 Jun 23. PMID 38913003
- [Derived] Shah SJ, Sharma K, Borlaug BA, Butler J, Davies M, Kitzman DW, Petrie MC, Verma S, Patel S, Chinnakondepalli KM, Einfeldt MN, Jensen TJ, Rasmussen S, Asleh R, Ben-Gal T, Kosiborod MN. Semaglutide and diuretic use in obesity-related heart failure with preserved ejection fraction: a pooled analysis of the STEP-HFpEF and STEP-HFpEF-DM trials. Eur Heart J. 2024 Sep 14;45(35):3254-3269. doi: 10.1093/eurheartj/ehae322. PMID 38739118
- [Derived] Butler J, Shah SJ, Petrie MC, Borlaug BA, Abildstrom SZ, Davies MJ, Hovingh GK, Kitzman DW, Moller DV, Verma S, Einfeldt MN, Lindegaard ML, Rasmussen S, Abhayaratna W, Ahmed FZ, Ben-Gal T, Chopra V, Ezekowitz JA, Fu M, Ito H, Lelonek M, Melenovsky V, Merkely B, Nunez J, Perna E, Schou M, Senni M, Sharma K, van der Meer P, Von Lewinski D, Wolf D, Kosiborod MN; STEP-HFpEF Trial Committees and Investigators. Semaglutide versus placebo in people with obesity-related heart failure with preserved ejection fraction: a pooled analysis of the STEP-HFpEF and STEP-HFpEF DM randomised trials. Lancet. 2024 Apr 27;403(10437):1635-1648. doi: 10.1016/S0140-6736(24)00469-0. Epub 2024 Apr 7. PMID 38599221
- [Derived] Kosiborod MN, Petrie MC, Borlaug BA, Butler J, Davies MJ, Hovingh GK, Kitzman DW, Moller DV, Treppendahl MB, Verma S, Jensen TJ, Liisberg K, Lindegaard ML, Abhayaratna W, Ahmed FZ, Ben-Gal T, Chopra V, Ezekowitz JA, Fu M, Ito H, Lelonek M, Melenovsky V, Merkely B, Nunez J, Perna E, Schou M, Senni M, Sharma K, van der Meer P, Von Lewinski D, Wolf D, Shah SJ; STEP-HFpEF DM Trial Committees and Investigators. Semaglutide in Patients with Obesity-Related Heart Failure and Type 2 Diabetes. N Engl J Med. 2024 Apr 18;390(15):1394-1407. doi: 10.1056/NEJMoa2313917. Epub 2024 Apr 6. PMID 38587233